CLINICAL TRIAL: NCT07029698
Title: Efficacy and Safety of a Parenterally Administered Fixed Vitamin Combination (Vitamin B6, B12 and Folic Acid) On Vitamin B12 Status and Methylation Capacity in Cobalamin Deficiency Compared to Oral Vitamin B12 Supplementation
Brief Title: A Study to See if a Combination of Vitamins That is Injected Into a Muscle is as Good and Safe as a Vitamin That is Taken by Mouth
Acronym: EASYVIT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6630-4200-42
Record Dates: First submitted 2025-05-01; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Vitamin B12 Deficiency
Keywords: Vitamin B12 deficiency; Vitamin B12 status; methylation capacity; holotranscobalamin; homocysteine; methylmalonic acid; folic acid; vitamin B6; S-adenosylmethione; S-adenosylhomocysteine
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12; Vitamin B 6; Folic Acid

STUDY DESIGN:
Intervention Model Description: This is a Phase IV, randomized, open label, controlled, multicenter, two parallel-group study in female and male patients with vitamin B12 deficiency, to assess the efficacy and safety of two different application routes of vitamin B12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin injection (Experimental): 1 injection twice weekly at the clinical site. Totally 8 injections through 4 week treatment period
  Interventions: Drug: Vitamin B12, Vitamin B6, Folic acid
- Vitamin B12 tablet (Active Comparator): 1 oral tablet once daily in the morning. Totally 28 tablets at approximately the same time each day through 4 week treatment period
  Interventions: Drug: Vitamin B12 (Cyanocobalamin)

INTERVENTIONS:
Drug: Vitamin B12, Vitamin B6, Folic acid — A solution for intramuscular injection of fixed vitamin combination (5 mg vitamin B6, 1 mg B12 and 1,05 mg folic acid )
  Other Names: Medivitan® iM
  Arms: Vitamin injection
Drug: Vitamin B12 (Cyanocobalamin) — oral tablets of 1mg Vitamin B12
  Other Names: B12 Ankermann®
  Arms: Vitamin B12 tablet

SUMMARY:
Primary efficacy objective:

To investigate the effects of a parenterally vitamin B12 combination treatment versus an oral vitamin B12 mono therapy on the vitamin B12 status in female and male patients as determined by the change from baseline in serum vitamin B12 concentration after 4 weeks (28 days) of treatment.

Secondary efficacy objectives:

To evaluate the effects of a parenterally vitamin B12 combination versus an oral vitamin B12 mono therapy after 4 weeks of treatment on:

* Serum holotranscobalamin
* Serum homocysteine
* Serum methylmalonic acid
* Combined vitamin B12 markers (cB12)
* Serum folic acid
* Serum vitamin B6
* Serum S-adenosylmethione (SAM)
* Serum S-adenosylhomocysteine (SAH)
* SAM/SAH ratio
* WHO-5 Well-Being Index
* Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36)
* Visual analogue scale (VAS) EQ-5D.

Safety objectives:

To evaluate the safety and tolerability of oral vitamin B12 mono therapy versus intramuscular vitamin B12 combination.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent to participate in the study (according to Order of the Ministry of Health of Ukraine No. 690 (with amendments)).
2. Female and male patients aged ≥18.
3. Vitamin B12 deficiency, defined as serum vitamin B12 < 350 pmol/L.
4. Female patients of childbearing potential (WOCBP) must be using two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc., with the exception of oral contraceptives), from the time of screening and for the duration of the study, through study completion and for 1 month following study completion. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Postmenopausal females must have had no regular menstrual bleeding for at least one (1) year prior to initial dosing. Female patients who report surgical sterilization must have had the procedure at least six (6) months prior to initial dosing. Surgical sterilization procedures should be supported with clinical documentation made available to the sponsor and noted in the Relevant Medical History / Current Medical Conditions section of the CRF. All female patients of childbearing potential must have negative pregnancy test results at screening. An additional pregnancy test will be performed on Days 0, 28, 56.
5. Able to communicate well with the investigator and able to understand and comply with the requirements of the study.
6. Patients are otherwise in relatively good health as determined by past medical history, physical examination, vital signs, and laboratory tests at screening (V -1).

Exclusion Criteria:

1. Active or recent vitamin B12, folic acid, B6 intake (the subject must not receive vitamin B12, folic acid, B6 drugs or food supplements for at least 6 months).
2. Participation in a previous clinical study with vitamin B12 within the 6 months prior to screening.
3. Any contraindication to one of the study drugs.
4. Pregnant or nursing (lactating) women.
5. Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
6. Subjects with anemia (hemoglobin < 10 mg/dL) or significant neurological symptoms due to vitamin B12 deficiency.
7. Any diseases that prevent intrinsic-factor independent passive diffusion in the small intestine (e.g. ileum resection)
8. Current drug addiction and/or alcohol abuse as evidenced by patient history and/or as determined by the investigator at V-1.
9. Cognitive or behavioural abnormalities that could impair the capacity to give informed consent or carry out protocol-specified procedures.
10. Inability to take oral medication.
11. Inability or unwillingness to comply with the study protocol.
12. Previous (last 6 months) or current participation in another clinical study.
13. Other medical, neuropsychiatric, or social conditions that, in the opinion of the investigator, are likely to adversely affect the risk-benefit of study participation, interfere with study compliance, or confound the study results.
14. Subjects who are in a dependent relationship with the Investigator or the Sponsor.
15. Subjects unwilling to give written informed consent to saving and/or propagation of anonymised medical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin B12 | Change from baseline at day 28
  Effects of treatment on serum vitamin B12

SECONDARY OUTCOMES:
Holotranscobalamin | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on serum holotranscobalamin
Homocystein | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on serum homocystein
Methylmalonic acid | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on serum methylmalonic acid
Combined vitamin B12 marker (cB12) | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on cB12. Combined vitamin B12 markers (cB12) will be statistically calculated using the levels of Serum holotranscobalamin, Serum homocysteine, Serum methylmalonic acid. cB12 (cB12=log10[(holoTC x B12)/(MMA x Hcy)]-(age factor).
Serum S-adenosylmethione (SAM) | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on serum S-adenosylmethione (SAM)
Serum S-adenosylhomocysteine (SAH) | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on serum S-adenosylhomocysteine (SAH)
SAM/SAH ratio | Change from baseline at day 28 and at follow up at day 56
  The change of the ratio will be assessed statistically using the levels of Serum S-adenosylmethione (SAM) and Serum S-adenosylhomocysteine (SAH)
Quality of life assessed with SF-36 | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on SF-36 questionnaire (from 0 to 100 points in each of the eight subscales, where the higher score means the higher quality of patient's life in each domain)
Quality of life assessed with WHO-5 questionnaire | Change from baseline at day 28 and at follow up at day 56
  Effects of treatment on WHO-5 questionnaire (from 0 to 25, where the higher score means the higher quality of patient's life)
Quality of life assessed with VAS EQ-5D | From baseline to day 28 and at follow up at day 56
  Effects of treatment on visual analogue scale EQ-5D (from 0 "the worst possible quality of life" to 10 "the best possible quality of life")

OTHER OUTCOMES:
Safety objectives | assessed through 56 days of patient's participation
  The evaluation of safety will be conducted through a comprehensive analysis of adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - State institution "V. Danilevsky Institute for Endocrine Pathology Problems of the NAMS of Ukraine", Kharkiv
  - Private Enterprise Private Manufacturing Company "Acinus", Kropyvnytskyi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Naurath HJ, Riezler R, Putter S, Ubbink JB. Does a single vitamin B-supplementation induce functional vitamin B-deficiency? Clin Chem Lab Med. 2001 Aug;39(8):768-71. doi: 10.1515/CCLM.2001.128. PMID 11592449
- [Background] Ubbink JB, van der Merwe A, Delport R, Allen RH, Stabler SP, Riezler R, Vermaak WJ. The effect of a subnormal vitamin B-6 status on homocysteine metabolism. J Clin Invest. 1996 Jul 1;98(1):177-84. doi: 10.1172/JCI118763. PMID 8690790
- [Background] Fedosov SN, Brito A, Miller JW, Green R, Allen LH. Combined indicator of vitamin B12 status: modification for missing biomarkers and folate status and recommendations for revised cut-points. Clin Chem Lab Med. 2015 Jul;53(8):1215-25. doi: 10.1515/cclm-2014-0818. PMID 25720072
- [Background] Metaxas C, Mathis D, Jeger C, Hersberger KE, Arnet I, Walter P. Early biomarker response and patient preferences to oral and intramuscular vitamin B12 substitution in primary care: a randomised parallel-group trial. Swiss Med Wkly. 2017 Apr 7;147:w14421. doi: 10.4414/smw.2017.14421. eCollection 2017. PMID 28421567
- [Background] Smith AD, Warren MJ, Refsum H. Vitamin B12. Adv Food Nutr Res. 2018;83:215-279. doi: 10.1016/bs.afnr.2017.11.005. Epub 2018 Feb 2. PMID 29477223
- [Background] Conzade R, Koenig W, Heier M, Schneider A, Grill E, Peters A, Thorand B. Prevalence and Predictors of Subclinical Micronutrient Deficiency in German Older Adults: Results from the Population-Based KORA-Age Study. Nutrients. 2017 Nov 23;9(12):1276. doi: 10.3390/nu9121276. PMID 29168737
- [Background] 1. Vitamin B12 (Cobalamine). Referenzwerte für die Nährstoffzufuhr. Bonn, Deutsche Gesellschaft für Ernährung, Österreichische Gesellschaft für Ernährung, Schweizerische Gesellschaft für Ernährung (Hrsg.). 4. Aktualisierte Ausgabe 2018.